CLINICAL TRIAL: NCT02544698
Title: Safety Study of Pneumococcal 13-valent Conjugate Vaccine in Healthy People Aged 2 Months and Older
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beijing Chaoyang District Centre for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: cycdc2015-2
Record Dates: First submitted 2015-09-06; First posted 2015-09-09 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2015-08

CONDITIONS: Pneumococcal 13-valent Conjugate Vaccine
Keywords: vaccine; safety

ARMS (4):
- One dose of PCV13a vaccine in aged 18 years and older (Experimental): One dose of PCV13a vaccine will be given in aged 18 years and older
  Interventions: Biological: One dose of PCV13a vaccine
- One dose of PCV13a vaccine in aged 2-5 years old (Experimental): One dose of PCV13a vaccine will be given in aged 2-5 years old
  Interventions: Biological: One dose of PCV13a vaccine
- One dose of PCV13 vaccine will be given at 2, 4, 6 months (Experimental): One dose of PCV13 vaccine will be given at 2, 4, 6 months respectively in aged 2 months old
  Interventions: Biological: three doses of PCV13a vaccine
- One dose of PCV13 vaccine will be given at 3、4、5 months (Experimental): One dose of PCV13 vaccine will be given at 3、4、5 months respectively in aged 3 months old
  Interventions: Biological: three doses of PCV13a vaccine

INTERVENTIONS:
Biological: One dose of PCV13a vaccine
  Arms: One dose of PCV13a vaccine in aged 18 years and older
Biological: One dose of PCV13a vaccine
  Arms: One dose of PCV13a vaccine in aged 2-5 years old
Biological: three doses of PCV13a vaccine
  Arms: One dose of PCV13 vaccine will be given at 2, 4, 6 months
Biological: three doses of PCV13a vaccine
  Arms: One dose of PCV13 vaccine will be given at 3、4、5 months

SUMMARY:
This study evaluates the safety of Pneumococcal 13-valent Conjugate Vaccine in Healthy People Aged 2 Months and Older.120 Subjects will be equally divided into 4 groups,including 18 years and older,2-5 years old, 2 months old and 3 months old. Subjects aged 18 years and 2-5 years old will receive one dose of PCV13 vaccine,while subjects aged 2 and 3 months will receive 3 doses of PCV13 vaccine,injected at 2, 4, 6 months or 3、4、5 months respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy babies with health conditions confirmed according to medical history, medical examination and judgment of researchers;
2. Satisfy the age requirements of the clinical trial.(children from 2 months to 5 years old and adults over the age of 18);
3. Parents or guardians of the subjects must provide informed consent forms with personally signature and date;
4. Parents or guardians of the subjects have been informed of all aspects of the research;
5. Subjects or guardians can obey the requirements of the clinical research;
6. No pneumococcal vaccine inoculation history, no other preventive vaccination within 7 days;
7. Axillary temperature below 37℃

Exclusion Criteria:

1. People with pneumococcal vaccine inoculation history, no matter experimentally or already on the market;
2. People has allergic reaction to any drugs, vaccine or vaccine-related components previously;
3. People has allergic reaction to 13vPnC, 7vPnC or other complexes associated with the drug, known or suspected;
4. People has hemorrhagic physical constitution or diseases that prolong bleeding time, intramuscular injection taboo;
5. People has immune deficiency or immune function inhibition, known or suspected;
6. People has irritability, convulsions, epilepsy, brain diseases and mental history or family history;
7. People has culture-confirmed invasive diseases caused by streptococcus pneumoniae history;
8. People has serious congenital malformations or serious chronic diseases that are known, people with congenital deformities, stunted or has a clinical diagnosis of serious chronic diseases (such as Down syndrome, diabetes, sickle cell anemia or nerve disorders, Guillain-Barre syndrome);
9. People suffers from these diseases: respiratory diseases, acute or chronic active stage of infection, severe cardiovascular disease, kidney and liver diseases, malignant tumors, skin diseases, babies with HIV infected mothers(inspection report is available);
10. People with vaccination-related contraindications that other researchers believe;
11. People take part in other clinical trials while taking part in this clinical trial or 28 days before this clinical trial. People who participate in purely observational studies are acceptable;
12. People received blood products or intravenous immunoglobulin. People who was inoculated Hepatitis B immunoglobulin can be acceptable.

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of adverse reactions of pneumococcal 13-valent conjugate vaccine | 3 months
  Adverse reactions associated with vaccine will be observed in subjects after vaccination. Solicited local adverse events include Pain, Redness, Swelling, Induration, Rash, Pruritus at injection site. solicited general adverse events include Fever, Nausea, Vomiting, Diarrhea, Decreased appetite, Be agitated (irritability, abnormal crying), fatigue, allergy